CLINICAL TRIAL: NCT01885494
Title: AFF008E:Observational Follow-up Extension Study to Evaluate Long-term Safety and Tolerability of Immunization With AFFITOPE® PD01A Applied During AFF008 in Patients With Parkinson's Disease.
Brief Title: AFF008E: Observational Phase 1b Follow-up Extension Study for Patients With Parkinson's Disease After Immunization With AFFITOPE® PD01A
Status: Completed | Type: Observational
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AFF008E; 2013-001774-20 (EudraCT Number)
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Analyzing patients' DNA (isolated out of whole blood) for polymorphisms in genes/regions like REP1 or alpha-synuclein to correlate results with the progression rate of the disease.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 15µg AFFITOPE® PD01A: Patients With Parkinson's Disease vaccinated with 4 injections of 15µg AFFITOPE® PD01A adsorbed to adjuvant during AFF008
- 75µg AFFITOPE® PD01A: Patients With Parkinson's Disease vaccinated with 4 injections of 75µg AFFITOPE® PD01A adsorbed to adjuvant during AFF008
- Control group: Untreated control group

SUMMARY:
AFF008E is set-up to assess the long term effects of the 4 PD01A vaccinations that have been applied during AFF008 with regard to safety as well as immunological-, radiological and clinical activity. Accordingly, during AFF008E, no further vaccine dose will be applied. Instead, patients who were participating in AFF008 will be assessed for another 52 weeks at the occasion of 4 quarterly visits. This is offered to patients who received PD01A vaccinations but also to the patients who served as controls in AFF008. Thus, AFF008E will ensure standardized and controlled management of individuals who have received PD01A as part of AFF008, the Phase I study analyzing for the first time in humans this first in class candidate.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated by the patient
* Participation in AFF008

Exclusion Criteria:

* History of questionable compliance to visit schedule; patients not expected to complete the clinical trial
* Participation in the active treatment phase of another clinical trial except AFF008 within 13 weeks before Visit 1 and for the whole study duration

Ages: 41 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only participants of AFF008 will be offered participation in AFF008E.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Tolerability and Safety | 52 weeks
  These will be based on the following parameters:
  * Withdrawal criteria (continuation decision) Number of patients who withdraw due to adverse events Reason for withdrawal
  * Occurrence of any serious adverse event possibly, probably or definitely related to the study vaccine at any time during the study.
  * Occurrence of any adverse events possibly, probably or definitely related to the study vaccine

SECONDARY OUTCOMES:
Immunological and Clinical Efficacy | 52 weeks
  Immunological parameters:
  -Titer of antibodies specific for the immunizing peptide, keyhole limpet hemocyanin (carrier protein), α-Synuclein, β-Synuclein as assessed by Enzyme-Linked Immunosorbent Assay
  Clinical efficacy variables:
  Motor symptoms:
  * Movement Disorder Society Unified Parkinson's Disease Rating Scale III
  * Investigator's Global Evaluation scale Non-motor symptoms
  * Parkinson's Disease Quality of Life-39 / Parkinson's Disease Non Motor Symptoms
  * Movement Disorder Society Unified Parkinson's Disease Rating Scale II
  * Cognitive scales
  * Smell identification test
  * Movement Disorder Society Unified Parkinson's Disease Rating Scale Ia (Caregiver-based assessment)
  * Geriatric Depression Scale Biomarker data
  * Change in Dopamine Transporter - Single Photon Emission Computed Tomography signal (compared to AFF008 results)
  * Assessment of change of volume of relevant brain regions (compared to AFF008 results)

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Volc, Prim. Dr., Principal Investigator — Studienzentrum der PROSENEX AmbulatoriumbetriebsgesmbH an der Confraternität-Privatklinik Josefstadt
Locations (1):
- Studienzentrum der PROSENEX, AmbulatoriumbetriebsgesmbH an der Confraternität-Privatklinik Josefstadt, Skodagasse 32, Vienna, Austria

REFERENCES:
- [Derived] McFarthing K, Simuni T. Clinical Trial Highlights: Targetting Alpha-Synuclein. J Parkinsons Dis. 2019;9(1):5-16. doi: 10.3233/JPD-189004. No abstract available. PMID 30741694